CLINICAL TRIAL: NCT02132039
Title: A Randomised Controlled Trial of Home-based Exercise Intervention for Caregivers of Persons With Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government); Chinese University of Hong Kong (Other); University of Melbourne (Other); National Ageing Research Institute, Australia (Other)
Responsible Party: Principal Investigator, Dr. Chan Wai Chi, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11121441
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Depression
Keywords: Tai Chi, dementia, caregivers
MeSH Terms: conditions — Depression; Dementia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12-step sitting Tai Chi Chuan (Active Comparator): The intervention is a simplified Tai Chi Chuan exercise, which consists of 12 steps, including weight shifting in different sitting positions, trunk and upper limb movements, and alternate thigh lift in a smooth and coordinated manner.
  Interventions: Other: 12-step sitting Tai Chi Chuan
- Control (Placebo Comparator): We provide participants in the control group with a level of social contact equivalent to the intervention group, which comprises structured conversations on topic other than physical activity.
  Interventions: Other: Control

INTERVENTIONS:
Other: 12-step sitting Tai Chi Chuan — The intervention consists of eight home-based sessions on 12-step sitting Tai Chi Chuan. Each session will last for an hour.
  Arms: 12-step sitting Tai Chi Chuan
Other: Control — The control consists of eight home-based sessions on useful health-care information. Each session will last for an hour.
  Arms: Control

SUMMARY:
The study aims to compare the efficacy of a home-based structured exercise programme (12-step sitting Tai Chi) involving both persons with dementia and their caregivers with a standard non-exercise social contact control in treating depression among caregivers. The effects of exercise on their cognition, quality of life and balance ability are also assessed. We will also examine if BDNF polymorphisms modulate mood changes in response to exercise intervention. Focus groups will be organised at the end to find out the facilitators and barriers in taking up exercise. The findings may offer an avenue of intervention by providing a low cost, relatively safe and effective treatment for dementia caregivers, which may in turn benefit the persons with dementia.

DETAILED DESCRIPTION:
The proposed study is a single-blind randomised controlled trial for two years. We will compare the efficacy of a home-based structured exercise programme (12-step sitting Tai Chi) for both carers and care recipients with a standard non-exercise social contact control in the treatment of depression among caregivers of persons with dementia. The study hypotheses include:

1. The structured home-based exercise programme will reduce caregiver depression. (Primary outcome)
2. The home-based exercise will improve caregivers' cognitive performance, quality of life and balance ability at the end of the study. (Secondary outcome)
3. The home-based exercise will improve the cognitive performance, quality of life and balance ability of persons with dementia at the end of the study. (Secondary outcome)
4. We also hypothesise that BDNF gene modulates mood changes in response to exercise intervention. (Secondary outcome)

ELIGIBILITY:
Inclusion Criteria:

Caregivers

* 18 years of age and above
* Live with persons with dementia
* 15-item Geriatric Depression Scale (GDS) >0 and <8
* No regular (i.e. ≥ 3 times/week) Tai Chi practice or other forms of mind-body exercise (e.g. yoga, qigong, mindfulness training) in the past six months
* Understand Chinese
* If they are on an antidepressant, they will not be included in the study unless they have been receiving pharmacological treatment on a steady dose for three months

Care recipient

* Aged 60 years or above
* Dementia diagnosis confirmed by a physician
* Dependence in at least one Activities of daily living(ADL)
* Mini Mental State Examination (MMSE) > 10
* No regular (i.e. ≥ 3 times/week) Tai Chi practice or other forms of mind-body exercise (e.g. yoga, qigong, mindfulness training) in the past six months

Exclusion Criteria:

Caregivers

* Presence of psychotic symptoms, imminently suicidal, unstable medical conditions (e.g. recent heart attack, recent stroke, episodes of dizziness, fainting attacks) or significant orthopaedic problems rendering participants unsuitable for physical training
* Carers who are found to have mental conditions that warrants psychiatric assessment and/or treatment (e.g. GDS >8, i.e. local cut-off score for significant depressive symptoms, or suicidal) will be referred to appropriate units for follow up

Care recipient

* Presence of psychotic symptoms, unstable medical conditions (e.g. recent heart attack, recent stroke, episodes of dizziness, fainting attacks) or significant orthopaedic problems rendering participants unsuitable for physical training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-09 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Hamilton Rating Scale for Depression in caregivers | Week 12
  The proportion of participants who are classified as responders by Hamilton Rating Scale for Depression (HAM-D-17). HAM-D-17 is a widely used and reliable measure of depressive symptoms. The scores range from 0 to 52, with higher scores indicating greater depression severity. Response to intervention is defined as a reduction of HAM-D-17 total score by ≥50% from baseline to endpoint.

SECONDARY OUTCOMES:
Berg Balance Scale in caregivers and care recipients | Week 12
  Berg Balance Scale (BBS)
Mini Mental State Examination in caregivers and care recipients | Week 12
  Global cognitive function will be measured by Mini Mental State examination (MMSE)
Quality of life in caregivers and care recipients | Week 12
  SF-12 Health Survey (SF-12)

CONTACTS AND LOCATIONS:
Overall Officials: Wai Chi Chan, Principal Investigator — The University of Hong Kong
Locations (5):
- China (5):
  - Hong Kong East Cluster, Hospital Authority, Hong Kong
  - Hong Kong West Cluster, Hospital Authority, Hong Kong
  - Kowloon West Cluster, Hospital Authority, Hong Kong
  - New Territories East Cluster, Hospital Authority, Hong Kong
  - New Territories West Cluster, Hospital Authority, Hong Kong

REFERENCES:
- [Derived] Chan WC, Lautenschlager N, Dow B, Ma SL, Wong CS, Lam LC. A home-based exercise intervention for caregivers of persons with dementia: study protocol for a randomised controlled trial. Trials. 2016 Sep 21;17(1):460. doi: 10.1186/s13063-016-1582-z. PMID 27655115